CLINICAL TRIAL: NCT00000439
Title: Efficacy of Valproate Maintenance in Bipolar Alcoholics
Brief Title: Drug Treatment for Alcoholics With Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAASAL10523
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Alcoholism; Bipolar Disorder
MeSH Terms: conditions — Alcoholism; Bipolar Disorder | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sodium valproate (Active Comparator): sodium valproate was added on treatment as usual and dose monitored by blood level measurements
  Interventions: Drug: sodium valproate
- placebo (Placebo Comparator): Placebo comparator was added on treatment as usual and dose monitored by blood level measurements
  Interventions: Drug: sodium valproate

INTERVENTIONS:
Drug: sodium valproate — subjects were randomized to sodium valproate vs placebo. Serum sodium valproate was monitored. This intervention was added on treatment as usual which was defined as being on lithium carbonate and also attending individual dual recovery counseling.
  Other Names: Depakote, Divalproex sodium, Depacon

SUMMARY:
The purpose of this study is to test the effectiveness of sodium valproate (Depacon) in treating individuals with alcohol dependence and comorbid bipolar disorder.

DETAILED DESCRIPTION:
The aim of this study is to test the mood stabilizer, anticonvulsant, sodium valproate in individuals with alcohol dependence and bipolar disorder, in a double-blind, placebo-controlled, and randomized trial of 6 months duration. All subjects are treated with treatment as usual, which include lithium carbonate and individual dual recovery counseling and are randomized to either sodium valproate or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Meets the criteria for alcohol dependence with comorbid bipolar disorder.
* Agreement to participate in outpatient treatment.
* Ability to tolerate lithium carbonate and be randomized to receive sodium valproate or placebo.
* Stable living situation.
* Ability to provide informed consent.

Exclusion Criteria:

* Psychiatric conditions including schizophrenia, schizoaffective disorder, any non-bipolar psychotic disorder, unipolar major depression, mental retardation, or signs of impaired cognitive functioning.
* Neurological conditions including epilepsy, history of brain injury, encephalitis, or any organic brain syndrome or focally abnormal electroencephalographic examination.
* Medical conditions including severe cardiac, liver, kidney, endocrine, hematologic, other impairing or unstable medical condition or impending surgery.
* Persistent elevation of liver function enzymes indicating active liver disease.
* Pregnancy or not using an acceptable contraceptive method.
* Inability to read or understand study forms; agree to informed consent.
* Impending incarceration or a mandate to attend treatment by the legal system for an alcohol use disorder.
* The presence of either/or cocaine dependence, opioid dependence, and intravenous drug use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2000-10; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Change in proportion of heavy drinking days | 6 months
  Change from baseline

SECONDARY OUTCOMES:
Changes in depressive and manic symptoms | 6 months
  Changes in depressive and manic symptoms scores from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ihsan M Salloum, MD, MPH, Principal Investigator — University of Miami
Locations (1):
- Department of Psychiatry, Western Psychiatric Institute and Clinic of the University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salloum IM, Cornelius JR, Daley DC, Kirisci L, Himmelhoch JM, Thase ME. Efficacy of valproate maintenance in patients with bipolar disorder and alcoholism: a double-blind placebo-controlled study. Arch Gen Psychiatry. 2005 Jan;62(1):37-45. doi: 10.1001/archpsyc.62.1.37. PMID 15630071